CLINICAL TRIAL: NCT04200105
Title: Endobronchial Ultrasound Transbronchial Needle Aspiration (EBUS-TBNA) Versus the Endobronchial Ultrasound Transbronchial Needle Biopsy Using the Acquire Needle in the Assessment of Mediastinal and Hilar Lymphadenopathy: a Randomised Trial
Brief Title: EBUS-TBNA vs Acquire TBNB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 274281
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Mediastinal Lymphadenopathy

STUDY DESIGN:
Intervention Model Description: 1:1 randomisation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EBUS TBNA (Active Comparator): Patients will undergo a standard EBUS examination, with sampling using a standard 22G EBUS needle.
  Interventions: Device: EBUS-TBNA
- Acquire TBNB (Experimental): Patients will undergo a standard EBUS examination, with sampling using an Acquire TBNB needle.
  Interventions: Device: Acquire TBNB

INTERVENTIONS:
Device: EBUS-TBNA — Mediastinal and hilar lymph node sampling using a standard 22G EBUS needle
  Arms: EBUS TBNA
Device: Acquire TBNB — Mediastinal and hilar lymph node sampling using the Acquire TBNB needle
  Arms: Acquire TBNB

SUMMARY:
This study aims to determine whether a new type of needle used for sampling lymph nodes (glands) around the airways of the lung, during a procedure called an endobronchial ultrasound (EBUS, provides more or better quality tissue to allow a definite diagnosis to be made than with the current standard sampling needle. Two hundred and fifty patients will be randomised to procedures using either the new or standard needle, and the results compared.

DETAILED DESCRIPTION:
The causes of mediastinal lymphadenopathy include infection, reactive lymphadenopathy, granulomatous disorders, and malignancy (metastases from various primaries, lymphoma, thymoma, neurogenic tumours). Radiological appearances are usually inadequate at providing a definitive diagnosis. In granulomatous disorders such as sarcoidosis as well as certain infections including tuberculosis, there is frequently mediastinal or hilar lymph node involvement without evidence of disease activity in other organs or lymph node groups. In malignancy, the metastatic involvement of lymph nodes has important prognostic significance. However, lymph node enlargement as seen on computerised tomography (CT) scanning is a poor predictor of disease involvement, and positron emission tomography (PET) of the mediastinum has a 10-15% false positive rate. Adequate mediastinal lymph node sampling is therefore essential in order to reach a definitive diagnosis and obtain satisfactory staging information.

Mediastinal nodal sampling has traditionally been performed using invasive surgical techniques which carry significant morbidity and mortality. These procedures (cervical mediastinoscopy, anterior mediastinotomy) require general anaesthesia and a hospital inpatient stay. Some patients with significant comorbidities are therefore not considered for these procedures as they are deemed unfit for anaesthesia. Safer, less invasive, and more cost-effective procedures using endoscopic ultrasonography to guide needle aspiration of mediastinal lymph nodes have been developed. Endobronchial ultrasound (EBUS) used to guide transbronchial needle aspiration (TBNA) of mediastinal masses has, in a matter of a few years, established itself firmly within the diagnostic and staging algorithm for lung cancer, and also in the diagnosis of other causes of mediastinal and hilar lymphadenopathy such as sarcoidosis and tuberculosis. A wide range of studies has demonstrated the effectiveness and safety of this technique, with various studies reporting sensitivities of between 67% and 92%3.

EBUS-guided needle aspirates performed with 22 gauge needles yield cytological specimens which are often inadequate at providing a firm diagnosis, or at confidently excluding other malignancies such as lymphoma. Immunohistochemistry and mutational analysis are today playing a more important role in the treatment of lung cancer. There is an increasing need for larger tissue samples and ideally biopsy material to enable advanced histopathological examination of specimens. For example, a substantial percentage of lung cancers express cell surface epidermal growth factor receptors (EGFRs). Small molecules designed to inhibit the tyrosine kinase (TK) domain of the EGFR, such as gefitinib and erlotinib, have demonstrated biologic and clinical responses in patients with mutations within the EGFR-TK domain. These TK inhibitors are now an important component of the armamentarium of the thoracic oncologist in the treatment of lung cancer. It has therefore become essential to establish the EGFR mutation status of lung cancers before consideration of treatment. Mutations of the KRAS gene in lung cancer patients have been shown to confer resistance to both erlotinib and gefitinib, adding to the importance of testing tissue samples for these mutations as well. In the past, tests for EGFR and KRAS gene mutations could only be performed on block tumours post resection, however advances in molecular biology in recent years have led to the ability to test small biopsy specimens for such mutations by polymerase chain reaction (PCR) analysis, fluorescence in situ hybridization (FISH) and immunohistochemistry (IHC). EBUS-TBNA, however, can only provide needle aspirates. These can provide samples adequate for cytological assessment, but do not always contain sufficient material to enable the formation of a cell block, thereby precluding histological assessment. Larger sized core tissue biopsy specimens are therefore likely to help in the histopathological assessment of lung cancer, and also in the diagnosis of sarcoidosis, lymphoma and other causes of mediastinal lymphadenopathy. This is likely to become even more important in the future as new clinically relevant genetic mutations are identified, and appropriate tests developed.

A novel transbronchial needle has been developed. This franseen needle has a crown tipped needle with three symmetrical cutting heels placed in a circumferential pattern designed with the intent to capture more tissue (figure 1). This needle tip was originally designed for use in interventional radiology, and is now the one of the leading designs used in endoscopic ultrasound of the gastrointestinal tract. This new needle can be passed down an EBUS scope and can hypothetically circumvent the deficiencies of EBUS-TBNA highlighted above by providing greater tissue volume for histological assessment and any subsequent molecular and genetic testing.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for EBUS-TBNA as part of clinical care
2. Lymph node size ≥5mm on CT scan
3. Age > 18 years
4. Written informed consent

Exclusion Criteria:

1. Contraindication to needle biopsy (e.g. coagulopathy, anticoagulation, thrombocytopenia, other bleeding diathesis)
2. Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-03-02 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
The difference in cell volume of cancer or other diagnostic tissue obtained between the two study arms | 1 week

SECONDARY OUTCOMES:
The difference between the two study arms in the percentage of lymph nodes sampled where enough tissue is obtained for complete immunohistochemical and genetic mutation analysis. | 1 month
The difference between the two study arms in the amount of DNA obtained. | 1 month
The difference in complication rates between the two study arms. | 1 month
The difference between the two study arms in yield (quantity of diagnostic material) in patients ultimately diagnosed with sarcoidosis. | 1 month
The difference between the two study arms in yield (quantity of diagnostic material) in patients ultimately diagnosed with lymphoma. | 1 month
The difference in sensitivity for detecting sarcoidosis between the two study arms. | 1 month
The difference in sensitivity for detecting lymphoma between the two study arms. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Samuel V Kemp, MBBS, Principal Investigator — Royal Brompton and Harefield NHS FT
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No